CLINICAL TRIAL: NCT06014216
Title: Treating Post-Operative Thirst With Flavoured Ice Lollies or Water - a Comparative Study to Improve Post-operative Discomfort
Acronym: THIRST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gloucestershire Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21/093/GHT
Record Dates: First submitted 2023-08-21; First posted 2023-08-28 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Postoperative Thirst
Keywords: Thirst; Postoperative; Ice Lollies; Anaesthesia; Hydration
MeSH Terms: interventions — Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients allocated ice lollies to treat post-operative thirst (Experimental): Ice lollies consisted of a flavoured ice popsicle (blackcurrant) provided through hospital catering. Participants were allocated a single ice popsicle with thirst scores recored pre and post intervention.
  Interventions: Other: Flavoured ice lollies (popsicles)
- Patients allocated water as control comparison (Other): Water is a routine treatment for post-operative thirst and therefore used a control to compare our intervention against.
  Interventions: Other: Water

INTERVENTIONS:
Other: Flavoured ice lollies (popsicles) — Blackcurrant flavoured ice popsicles, 105ml volume.
  Arms: Patients allocated ice lollies to treat post-operative thirst
Other: Water — Water from tap, one cup given by recovery nurses.
  Arms: Patients allocated water as control comparison

SUMMARY:
Patients are asked not to eat and drink before their operation, and we know that this can make people feel thirstier when they wake up from their anaesthetic. We want to know if giving patients ice lollies improves their thirst more than if they were given water. Gloucestershire Royal Hospital is funding and running a research study to find ways to try and improve this.

DETAILED DESCRIPTION:
The 2019 peri-operative quality improvement project (PQIP) run by the Royal College of Anaesthetists showed 79% of patients experience moderate to severe thirst post-operatively. As a significant source of post-operative discomfort, resolving patient thirst may significantly improve their experience.

Whilst provision of oral fluids may be able to alleviate some thirst, many patients are unable to drink sufficient quantities to quench their thirst following an anaesthetic. Furthermore, studies have shown that frozen water is able to quench thirst to a greater degree than liquids.

The purpose of this study is to determine whether ice lollies quench post-operative thirst to a greater degree than water. Patients are already routinely offered water post-operatively, the offering of flavoured ice lollies is a novel intervention for our hospital. We intend to investigate two primary outcomes. First, can ice lollies quench post-operative thirst to a greater degree than water and therefore improve patient discomfort. Second, if ice lollies are found to be superior to water in quenching thirst and improving post-operative discomfort, do these patients take less time to recover from their operation?

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 18 years of age
2. Patients attending for elective surgery

Exclusion Criteria:

1. Allergy to products within the ice lolly
2. Designated nil-by-mouth by anaesthetic or surgical teams
3. Patient less than 18 years old
4. Patient unable to give consent
5. Refusal of patient to be involved with study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2021-05-17 (Actual); Study Completion 2021-05-17 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is the level of post-operative thirst following intervention with either water or ice lolly. | Intervention is to be given when the patient is adequately recovered from anaesthesia. An initial thirst score is recorded, then intervention given. Thirst scores are recorded again 15 minutes later to provide data for the primary outcome measure.
  Data on pre and post-intervention thirst will be recorded using questionnaires and a numerical rating score from 0 to 10, with 0 being no thirst at all and 10 being very thirsty. These scores will also be sub-divided into no thirst (0), mild thirst (1-3), moderate thirst (4-7) and severe thirst (8-10). This data will undergo statistical analysis to challenge the null hypothesis for the primary outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: David Sleep, BSc MSc MBBS D.Phil, Principal Investigator — Gloucestershire Hospitals NHS Foundation Trust
Locations (1):
- Gloucestershire Royal Hospital, Gloucester, Gloucestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
This is a small centre study with a minor intervention. Participant information is limited to demographic and operative data only.